CLINICAL TRIAL: NCT02258139
Title: The Study to Evaluate the Product Performance of a New Silicone Hydrogel Contact Lens
Brief Title: Study to Evaluate the Product Performance of a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-002
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Corneal Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group 1 (Experimental): 1st overnight visit with no contact lens; 2nd overnight visit randomized to either left or right eye for B&L Investigational Contact Lens
  Interventions: Device: B&L Investigational Contact Lens

INTERVENTIONS:
Device: B&L Investigational Contact Lens — The lens used in this study will be supplied by the Sponsor. All subjects will wear a -3.00D lens.

SUMMARY:
This will be a randomized non-dispensing study comparing the overnight corneal swelling of an eye while wearing no contact lens to the Ultra contract lens.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 40 years of age (inclusive)
* Not a current contact lens wearer (have not worn extended wear, and not worn in lenses in 6 months)
* Able to read, comprehend and sign an informed consent
* Willing to comply with the wear and study visit schedule
* Monocular best-corrected distance visual acuity >/-20/25 in each eye

Exclusion Criteria:

* Any active corneal infection, disease, injury, inflammation, past surgery, or ocular abnormality which may interfere with contact lens wear
* Systemic or ocular allergies, which might interfere with contact lens wear
* Systemic disease or condition, which might interfere with contact lens wear
* Use of prescription sleep aids or alcohol within 24 hours of study appointment
* Inability to wear contact lenses
* Under 18 years of age

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2014-12-11 (Actual); Study Completion 2014-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, OD, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Indiana University, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group 1
Started | 38
Completed | 30
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Study Group 1
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Central Corneal Thickness
Description: Percent change in central corneal thickness from evening to morning (after 8 hours with lid closed)
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Study Group 1
Number analyzed (Participants) | 38
milimeters
  Visit 1 (without lens) | 4.01 (1.57)
  Visit 2 (with lens) | 5.57 (2.11)

2. Secondary Outcome: Time to Restore Central Corneal Thickness
Description: Time (hours) to restore central corneal thickness to its baseline value after lens removal
Time Frame: 48 hours
Measure: Number; unit: percentage of participants
Groups:
- Test Eye With Lens: Test eye after lens removed
- Control Eye: Control eye in subjects with lens in test eye
Arm/Group | Test Eye With Lens | Control Eye
Number analyzed (Participants) | 38 | 38
percentage of participants
  0 hours | 0 | 5.3
  1 hours | 34.2 | 63.2
  2 hours | 44.7 | 23.7
  3 hours | 15.8 | 5.3
  4 hours | 5.3 | 2.6
  >4 hours | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable.
Arm/Group | Study Group 1
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.